CLINICAL TRIAL: NCT02296125
Title: A Phase III, Double-blind, Randomised Study to Assess the Safety and Efficacy of AZD9291 Versus a Standard of Care Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor as First Line Treatment in Patients With Epidermal Growth Factor Receptor Mutation Positive, Locally Advanced or Metastatic Non Small Cell Lung Cancer.
Brief Title: AZD9291 Versus Gefitinib or Erlotinib in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Acronym: FLAURA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5160C00007; U1111-1160-2242 (Other Grant/Funding Number: 112455); 2014-002694-11 (EudraCT Number)
Record Dates: First submitted 2014-10-22; First posted 2014-11-20 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced or Metastatic EGFR Sensitising Mutation Positive Non Small Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer; EGFRm+; AZD9291; TKI; Phase III
MeSH Terms: interventions — osimertinib; Erlotinib Hydrochloride; Gefitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZD9291+ placebo (Experimental): AZD9291 (80 mg or 40 mg orally, once daily) plus placebo Erlotinib (150mg or 100mg orally, once daily) or placebo Gefitinib (250 mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: AZD9291 80 mg/40 mg + placebo; Drug: Placebo Erlotinib 150/100mg; Drug: Placebo Gefitinib 250 mg
- Standard of Care + placebo AZD9291 (Active Comparator): Erlotinib (150 mg or 100 mg orally, once daily) or placebo Gefitinib (250 mg orally, once daily) plus placebo AZD9291 (80 mg or 40 mg orally, once daily), in accordance with the randomisation schedule.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Standard of Care arm may have the option to receive open-label AZD9291 (crossover to active AZD9291).
  Interventions: Drug: Erlotinib 150/100 mg; Drug: Gefitinib 250 mg; Drug: Placebo AZD9291 80 mg/ 40 mg

INTERVENTIONS:
Drug: AZD9291 80 mg/40 mg + placebo — The initial dose of AZD9291 80 mg once daily can be reduced to 40 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: AZD9291+ placebo
Drug: Placebo Erlotinib 150/100mg — The initial dose of Placebo Erlotinib 150 mg once daily can be reduced to Placebo 100 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Placebo Tarceva 150/100 mg
  Arms: AZD9291+ placebo
Drug: Placebo Gefitinib 250 mg — The initial dose of Placebo Gefitinib 250 mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Placebo Iressa 250 mg
  Arms: AZD9291+ placebo
Drug: Erlotinib 150/100 mg — The initial dose of Erlotinib 150mg once daily can be reduced to 10 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Standard of Care arm may have the option to receive open-label AZD9291 (crossover to active AZD9291).
  Other Names: Tarceva 150/100 mg
  Arms: Standard of Care + placebo AZD9291
Drug: Gefitinib 250 mg — The initial dose of Gefitinib 250mg once daily cannot be reduced. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Following objective disease progression according to RECIST 1.1, as per investigator assessment, patients who were randomized to Standard of Care arm may have the option to receive open-label AZD9291 (crossover to active AZD9291).
  Other Names: Iressa 250mg
  Arms: Standard of Care + placebo AZD9291
Drug: Placebo AZD9291 80 mg/ 40 mg — The initial dose of Placebo AZD9291 80 mg once daily can be reduced to Placebo AZD9291 40 mg once daily under specific circumstances. A cycle of treatment is defined as 21 days of once daily treatment. Number of cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Arms: Standard of Care + placebo AZD9291

SUMMARY:
To assess the efficacy and safety of AZD9291 versus a standard of care epidermal growth factor receptor tyrosine kinase inhibitor in patients with locally advanced or Metastatic Non Small Cell Lung Cancer

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomised study assessing the efficacy and safety of AZD9291 (80 mg orally, once daily) versus a standard of care (SoC) Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) (either gefitinib [250 mg orally, once daily] or erlotinib [150 mg orally, once daily]) in patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) that is known to be EGFR sensitising mutation (EGFRm) positive, treatment-naïve and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged at least 18 years.
2. Pathologically confirmed adenocarcinoma of the lung.
3. Locally advanced or metastatic NSCLC, not amenable to curative surgery or radiotherapy.
4. The tumour harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R).
5. Mandatory provision of an unstained, archived tumour tissue sample in a quantity sufficient to allow for central analysis of EGFR mutation status.
6. Patients must be treatment-naïve for locally advanced or metastatic NSCLC and eligible to receive first-line treatment with gefitinib or erlotinib as selected by the participating centre. Prior adjuvant and neo-adjuvant therapy is permitted(chemotherapy, radiotherapy, investigational agents).
7. Provision of informed consent prior to any study specific procedures, sampling, and analysis.
8. World Health Organization Performance Status of 0 to 1 with no clinically significant deterioration over the previous 2 weeks and a minimum life expectancy of 12 weeks

Exclusion Criteria:

1. Treatment with any of the following:

   * Prior treatment with any systemic anti-cancer therapy for locally advanced/metastatic NSCLC.
   * Prior treatment with an EGFR-TKI.
   * Major surgery within 4 weeks of the first dose of study drug.
   * Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug.
   * Patients currently receiving medications or herbal supplements known to be potent inducers of cytochrome P450 (CYP) 3A4.
   * Alternative anti-cancer treatment
   * Treatment with an investigational drug within five half-lives of the compound or any of its related material.
2. Any concurrent and/or other active malignancy that has required treatment within 2 years of first dose of study drug.
3. Spinal cord compression, symptomatic and unstable brain metastases, except for those patients who have completed definitive therapy, are not on steroids, have a stable neurologic status for at least 2 weeks after completion of the definitive therapy and steroids.
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses; or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV).
5. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product, or previous significant bowel resection that would preclude adequate absorption of AZD9291.
6. Any of the following cardiac criteria:

   * Mean resting corrected QT interval (QTc) >470 msec, obtained from 3 ECGs, using the screening clinic ECG machine-derived QTcF value.
   * Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG.
   * Any patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
7. Past medical history of ILD, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
8. Involvement in the planning and/or conduct of the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Actual)
Dates: Start 2014-12-03 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2025-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (147):
- United States (13):
  - Research Site, Anaheim, California
  - Research Site, Santa Rosa, California
  - Research Site, West Hills, California
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Louisville, Kentucky
  - Research Site, Bethesda, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Lebanon, New Hampshire
  - Research Site, Salisbury, North Carolina
  - Research Site, Burlington, Vermont
- Australia (7):
  - Research Site, Camperdown
  - Research Site, Chermside
  - Research Site, Clayton
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, Nedlands
  - Research Site, Woolloongabba
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Roeselare
- Research Site, Porto Alegre, Brazil
- Research Site, Sofia, Bulgaria
- Canada (4):
  - Research Site, Edmonton, Alberta
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- China (15):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Suzhou
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yangzhou
- Research Site, Ostrava, Czechia
- France (6):
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Lyon
  - Research Site, Nantes
  - Research Site, Toulon Naval
  - Research Site, Villejuif
- Germany (9):
  - Research Site, Bad Berka
  - Research Site, Berlin
  - Research Site, Gauting
  - Research Site, Halle
  - Research Site, Heidelberg
  - Research Site, Karlsruhe
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Villingen-Schwenningen
- Hungary (6):
  - Research Site, Farkasgyepü
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Miskolc
  - Research Site, Székesfehérvár
  - Research Site, Tatabánya
  - Research Site, Zalaegerszeg
- Israel (4):
  - Research Site, Haifa
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Tel Litwinsky
- Italy (8):
  - Research Site, Cremona
  - Research Site, Lecce
  - Research Site, Lecco
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Roma
  - Research Site, Sondrio
  - Research Site, Terni
- Japan (15):
  - Research Site, Chūōku
  - Research Site, Fukuoka
  - Research Site, Hirakata-shi
  - Research Site, Kanazawa
  - Research Site, Kashiwa
  - Research Site, Kobe
  - Research Site, Matsuyama
  - Research Site, Natori-shi
  - Research Site, Osaka
  - Research Site, Osakasayama-shi
  - Research Site, Sagamihara-shi
  - Research Site, Sakaishi
  - Research Site, Sendai
  - Research Site, Sunto-gun
  - Research Site, Yokohama
- Malaysia (3):
  - Research Site, Kuala Lumpur
  - Research Site, Kuantan
  - Research Site, Kuching
- Philippines (3):
  - Research Site, Cebu
  - Research Site, Manila
  - Research Site, Quezon City
- Poland (5):
  - Research Site, Brzozoów
  - Research Site, Otwock
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Warsaw
- Portugal (4):
  - Research Site, Amadora
  - Research Site, Lisbon
  - Research Site, Porto
  - Research Site, Vila Nova de Gaia
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Craiova
- Research Site, Saint Petersburg, Russia
- South Korea (4):
  - Research Site, Cheongju-si
  - Research Site, Incheon
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Lleida
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Seville
  - Research Site, Zaragoza
- Research Site, Linköping, Sweden
- Switzerland (3):
  - Research Site, Lucerne
  - Research Site, Winterthur
  - Research Site, Zurich
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taoyuan
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Muang
- Turkey (Türkiye) (3):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- Ukraine (4):
  - Research Site, Dnipro
  - Research Site, Kryvyi Rih
  - Research Site, Lviv
  - Research Site, Sumy
- United Kingdom (4):
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Maidstone
  - Research Site, Withington
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Markovets A, Merino Vega D, Abbosh C, Quinn K, Chang K, Wienke S, Hartmaier R, Barrett JC, Hodgson D. Variability of Circulating Tumor DNA Levels in Plasma Samples From Patients With Advanced Non-Small-Cell Lung Cancer in the Absence of Treatment. JCO Precis Oncol. 2025 Oct;9:e2500287. doi: 10.1200/PO-25-00287. Epub 2025 Oct 30. PMID 41166679
- [Derived] Murat-Onana ML, Ramalingam SS, Janne PA, Gray JE, Ahn MJ, John T, Yatabe Y, Huang X, Rukazenkov Y, Javey M, Brown H, Li-Sucholeiki X. EGFR mutation testing across the osimertinib clinical program. Lung Cancer. 2025 Jun;204:108549. doi: 10.1016/j.lungcan.2025.108549. Epub 2025 Apr 18. PMID 40311309
- [Derived] Viray H, Piper-Vallillo AJ, Widick P, Academia E, Shea M, Rangachari D, VanderLaan PA, Kobayashi SS, Costa DB. A Real-World Study of Patient Characteristics and Clinical Outcomes in EGFR Mutated Lung Cancer Treated with First-Line Osimertinib: Expanding the FLAURA Trial Results into Routine Clinical Practice. Cancers (Basel). 2024 Mar 7;16(6):1079. doi: 10.3390/cancers16061079. PMID 38539415
- [Derived] Johnson M, Serra Traynor C, Vishwanathan K, Overend P, Hartmaier R, Markovets A, Chmielecki J, Mugundu GM, Barrett JC, Tomkinson H, Ramalingam SS. Longitudinal Circulating Tumor DNA Modeling to Predict Disease Progression in First-Line Mutant Epidermal Growth Factor Receptor Non-Small Cell Lung Cancer. Clin Pharmacol Ther. 2024 Feb;115(2):349-360. doi: 10.1002/cpt.3113. Epub 2023 Dec 21. PMID 38010260
- [Derived] Walding A, Skaltsa K, Casamayor M, Ryden A. Time to deterioration of patient-reported outcomes in non-small cell lung cancer: exploring different definitions. Qual Life Res. 2022 Aug;31(8):2535-2543. doi: 10.1007/s11136-022-03088-0. Epub 2022 Jan 31. PMID 35099678
- [Derived] Cheng Y, He Y, Li W, Zhang HL, Zhou Q, Wang B, Liu C, Walding A, Saggese M, Huang X, Fan M, Wang J, Ramalingam SS. Osimertinib Versus Comparator EGFR TKI as First-Line Treatment for EGFR-Mutated Advanced NSCLC: FLAURA China, A Randomized Study. Target Oncol. 2021 Mar;16(2):165-176. doi: 10.1007/s11523-021-00794-6. Epub 2021 Feb 5. PMID 33544337
- [Derived] Leighl NB, Karaseva N, Nakagawa K, Cho BC, Gray JE, Hovey T, Walding A, Ryden A, Novello S. Patient-reported outcomes from FLAURA: Osimertinib versus erlotinib or gefitinib in patients with EGFR-mutated advanced non-small-cell lung cancer. Eur J Cancer. 2020 Jan;125:49-57. doi: 10.1016/j.ejca.2019.11.006. Epub 2019 Dec 12. PMID 31838405
- [Derived] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Derived] Brown H, Vansteenkiste J, Nakagawa K, Cobo M, John T, Barker C, Kohlmann A, Todd A, Saggese M, Chmielecki J, Markovets A, Scott M, Ramalingam SS. Programmed Cell Death Ligand 1 Expression in Untreated EGFR Mutated Advanced NSCLC and Response to Osimertinib Versus Comparator in FLAURA. J Thorac Oncol. 2020 Jan;15(1):138-143. doi: 10.1016/j.jtho.2019.09.009. Epub 2019 Oct 9. PMID 31605792
- [Derived] Gray JE, Okamoto I, Sriuranpong V, Vansteenkiste J, Imamura F, Lee JS, Pang YK, Cobo M, Kasahara K, Cheng Y, Nogami N, Cho EK, Su WC, Zhang G, Huang X, Li-Sucholeiki X, Lentrichia B, Dearden S, Jenkins S, Saggese M, Rukazenkov Y, Ramalingam SS. Tissue and Plasma EGFR Mutation Analysis in the FLAURA Trial: Osimertinib versus Comparator EGFR Tyrosine Kinase Inhibitor as First-Line Treatment in Patients with EGFR-Mutated Advanced Non-Small Cell Lung Cancer. Clin Cancer Res. 2019 Nov 15;25(22):6644-6652. doi: 10.1158/1078-0432.CCR-19-1126. Epub 2019 Aug 22. PMID 31439584
- [Derived] Planchard D, Boyer MJ, Lee JS, Dechaphunkul A, Cheema PK, Takahashi T, Gray JE, Tiseo M, Ramalingam SS, Todd A, McKeown A, Rukazenkov Y, Ohe Y. Postprogression Outcomes for Osimertinib versus Standard-of-Care EGFR-TKI in Patients with Previously Untreated EGFR-mutated Advanced Non-Small Cell Lung Cancer. Clin Cancer Res. 2019 Apr 1;25(7):2058-2063. doi: 10.1158/1078-0432.CCR-18-3325. Epub 2019 Jan 18. PMID 30659024
- [Derived] Ohe Y, Imamura F, Nogami N, Okamoto I, Kurata T, Kato T, Sugawara S, Ramalingam SS, Uchida H, Hodge R, Vowler SL, Walding A, Nakagawa K. Osimertinib versus standard-of-care EGFR-TKI as first-line treatment for EGFRm advanced NSCLC: FLAURA Japanese subset. Jpn J Clin Oncol. 2019 Jan 1;49(1):29-36. doi: 10.1093/jjco/hyy179. PMID 30508196
- [Derived] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- See also: Cancer — http://www.nlm.nih.gov/medlineplus/cancer.html
- See also: Lung Cancer — http://www.nlm.nih.gov/medlineplus/lungcancer.html
- See also: Erlotinib — http://druginfo.nlm.nih.gov/drugportal/ProxyServlet?mergeData=true&objectHandle=DBMaint&APPLICATION_NAME=drugportal&actionHandle=default&nextPage=jsp/drugportal/ResultScreen.jsp&TXTSUPERLISTID=0183321746&QV1=ERLOTINIB
- See also: FDA Drug and Device Resources — https://clinicaltrials.gov/ct2/info/fdalinks
- See also: Gefitinib — http://www.fda.gov/Drugs/DrugSafety/PostmarketDrugSafetyInformationforPatientsandProviders/ucm110473.htm
- See also: EGFR mutation — http://vsearch.nlm.nih.gov/vivisimo/cgi-bin/query-meta?v%3Aproject=medlineplus&query=EGFR+mutation&x=20&y=19
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3062&filename=FLAURA_Redacted.pdf
- See also: Clinical Study Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3062&filename=Final%20to%20Client_D5160C00007_CSP_A.pdf
- See also: SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3062&filename=Final%20to%20Client_D5160C00007_SAP_A.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 556 participants in Global cohort (out of 673 participants in Global and China cohorts) were randomized to treatment at 132 study centres in 29 countries. An additional 117 participants in 19 centres were enrolled into the China extension cohort only.
Pre-assignment Details: During the 28 day screening period, participants were enrolled based on the presence in their tumour of at least 1 of the 2 most frequent Epidermal growth factor receptor (EGFR) mutations. At the time of enrolment, all participants were required to provide biopsy tissue for central testing of the Exon 19 deletion (Ex19del) and L858R mutations
Groups:
- Osimertinib 80 mg (Global Cohort); Osimertinib 80 mg (China Cohort): Randomized participants received Osimertinib 80 mg orally once daily (QD)
- SoC EGFR-TKI (Global Cohort): Randomized participant received Standard of care (SoC) Epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI). Participants received gefitinib 250 mg orally QD or erlotinib 150 mg orally QD.
- SoC EGFR-TKI (China Cohort): Randomized participant received Standard of care (SoC) Epidermal growth factor receptor-tyrosine kinase inhibitor (EGFRTKI). Participants received gefitinib 250 mg orally QD or erlotinib 150 mg orally QD.
Period: Overall Study
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Started (There were 19 participants double counted which shows the total participants of 692.) | 279 | 277 (183 participant received gefitinib and 93 participants received erlotinib.) | 71 (There were 12 participants who were in both the Global and China Extension Osimertinib Arm.) | 65 (There were 7 participants who were in both the Global and China Extension SoC EGFR-TKI Arm.)
Completed (Participants ongoing study treatment at data cut-off) | 61 | 13 | 15 | 3
Not Completed | 218 | 264 | 56 | 62
Not completed — Withdrawal by Subject | 18 | 8 | 6 | 2
Not completed — Adverse Event | 41 | 52 | 9 | 4
Not completed — Severe non-compliance to protocol | 0 | 1 | 0 | 0
Not completed — Condition under investigation worsened | 153 | 199 | 39 | 56
Not completed — Any reason not specifically recorded | 6 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: There were 12 participants who were in both the Global and China Extension Osimertinib Arm and 7 participants in both the Global and China Extension SoC EGFR-TKI arm.
Groups:
- Global + China Extension Osimertinib Arm: All participants who were enrolled in Osimertinib Arm for either the global or China Extension study.
- Global + China Extension SoC EGFR-TKI Arm: All participants who were enrolled in SoC EGFR-TKI Arm for either the Global or China Extension study
- Total: Total of all reporting groups
Arm/Group | Global + China Extension Osimertinib Arm | Global + China Extension SoC EGFR-TKI Arm | Total
Number analyzed (Participants) | 338 | 335 | 673
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Each study is reported in a seprate row. There were 12 participants who were in both the Global and China Extension Osimertinib Arm, and 7 particicpants in both the Global and China Extension SoC EGFR-TKI arm.
  Years
    Global cohort: number analyzed (Participants) | 279 | 277 | 556
    Global cohort | 62.7 (10.70) | 63.3 (10.90) | 63.0 (10.79)
    China Cohort: number analyzed (Participants) | 71 | 65 | 136
    China Cohort | 59.1 (9.66) | 59.0 (10.94) | 59.0 (10.26)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Each study is reported in a seprate row. There were 12 participants who were in both the Global and China Extension Osimertinib Arm, and 7 particicpants in both the Global and China Extension SoC EGFR-TKI arm.
  Participants
    Global cohort: number analyzed (Participants) | 279 | 277 | 556
    Global cohort: Female | 178 | 172 | 350
    Global cohort: Male | 101 | 105 | 206
    China Cohort: number analyzed (Participants) | 71 | 65 | 136
    China Cohort: Female | 43 | 46 | 89
    China Cohort: Male | 28 | 19 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Each study is reported in a seprate row. There were 12 participants who were in both the Global and China Extension Osimertinib Arm, and 7 particicpants in both the Global and China Extension SoC EGFR-TKI arm.
  Participants
    Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Global Cohort: American Indian or Alaska Native | 1 | 1 | 2
    Global Cohort: Asian | 174 | 173 | 347
    Global Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Global Cohort: Black or African American | 2 | 2 | 4
    Global Cohort: White | 101 | 100 | 201
    Global Cohort: More than one race | 0 | 0 | 0
    Global Cohort: Unknown or Not Reported | 1 | 1 | 2
    China Cohort: number analyzed (Participants) | 71 | 65 | 136
    China Cohort: American Indian or Alaska Native | 0 | 0 | 0
    China Cohort: Asian | 71 | 65 | 136
    China Cohort: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    China Cohort: Black or African American | 0 | 0 | 0
    China Cohort: White | 0 | 0 | 0
    China Cohort: More than one race | 0 | 0 | 0
    China Cohort: Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Each study is reported in a seprate row. There were 12 participants who were in both the Global and China Extension Osimertinib Arm, and 7 particicpants in both the Global and China Extension SoC EGFR-TKI arm.
  Participants
    Asian-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Asian-Global Cohort | 77 | 94 | 171
    Chinese-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Chinese-Global Cohort | 32 | 24 | 56
    Japanese-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Japanese-Global Cohort | 65 | 55 | 120
    Other-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Other-Global Cohort | 103 | 104 | 207
    Missing-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Missing-Global Cohort | 2 | 0 | 2
    Hispanic or Latino-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Hispanic or Latino-Global Cohort | 0 | 0 | 0
    Chinese-China cohort: number analyzed (Participants) | 71 | 65 | 136
    Chinese-China cohort | 71 | 65 | 136
Smoking status [Count of Participants; unit: Participants] — Population: Each study is reported in a seprate row. There were 12 participants who were in both the Global and China Extension Osimertinib Arm, and 7 particicpants in both the Global and China Extension SoC EGFR-TKI arm.
  Participants
    Never smoked-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Never smoked-Global Cohort | 182 | 175 | 357
    Current smokers-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Current smokers-Global Cohort | 8 | 9 | 17
    Former smokers-Global Cohort: number analyzed (Participants) | 279 | 277 | 556
    Former smokers-Global Cohort | 89 | 93 | 182
    Never smoked-China Cohort: number analyzed (Participants) | 71 | 65 | 136
    Never smoked-China Cohort | 53 | 50 | 103
    Current smokers-China Cohort: number analyzed (Participants) | 71 | 65 | 136
    Current smokers-China Cohort | 3 | 4 | 7
    Former smokers-China Cohort: number analyzed (Participants) | 71 | 65 | 136
    Former smokers-China Cohort | 15 | 11 | 26

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS) (Months)
Description: Progression-free survival was defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression and was used to assess the efficacy of single agent osimertinib compared with SoC EGFR-TKI therapy as measured by PFS. The primary endpoint of PFS was based on Investigator assessment.
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks relative to randomisation until progression
Population: The full analysis set (FAS) and China-only FAS. FAS included all randomized participants prior to the end of global recruitment. The China-only FAS included all China participants randomized in mainland-China as part of the global study and all additional China participants recruited in mainland China after global recruitment was completed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Months | 18.9 [15.2 to 21.4] | 10.2 [9.6 to 11.1] | 17.8 [13.6 to 20.7] | 9.8 [8.3 to 13.8]
Statistical Analysis 1: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.37 to 0.57]
Statistical Analysis 2: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.0065, Log Rank; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.37 to 0.85]

2. Primary Outcome: Percentage of Participants in Progression Free Survival at 6, 12, and 18 Months
Description: Progression-free survival was defined as the time from randomization until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the participant withdrew from randomized therapy or received another anti-cancer therapy prior to progression and was used to assess the efficacy of single agent osimertinib compared with SoC EGFR-TKI therapy as measured by PFS.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Percentage of Participants
  Progression free at 6 months (%) | 88.4 | 75.2 | 78.8 | 72.3
  Progression free at 12 months (%) | 68.2 | 42.3 | 67.3 | 44.6
  Progression free at 18 months (%) | 50.9 | 24.4 | 46.9 | 25.8

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the number (%) of participants with measurable disease with at least 1 visit response of Complete response (CR) or Partial response (PR) and it was used to further assess the efficacy of osimertinib compared with SoC EGFR-TKI therapy. ORR was based on Investigator assessment.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Percentage of participants | 76.7 [71.29 to 81.53] | 69.0 [63.14 to 74.35] | 76.1 [64.5 to 85.4] | 70.8 [58.2 to 81.4]
Statistical Analysis 1: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p = 0.036, Regression, Logistic; Odds Ratio (OR) = 1.51, 95% CI 2-sided [1.03 to 2.22]
Statistical Analysis 2: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.485, Regression, Logistic; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.61 to 2.84]

4. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response was defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression and was used to further assess the efficacy of osimertinib compared with SoC EGFR-TKI therapy.
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks until objective disease progression
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Months | 17.2 [13.8 to 22.0] | 8.5 [7.3 to 9.8] | 16.4 [12.3 to NA] — NA-Upper limit is not calculable at this data cut-off. | 10.9 [8.3 to 13.8]
Statistical Analysis 1: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.0133, Regression, Linear; Mean Difference (Final Values) = 2.48, 95% CI 2-sided [1.21 to 5.09]
Statistical Analysis 2: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p < 0.0001, Regression, Linear; Mean Difference (Final Values) = 2.27, 95% CI 2-sided [1.68 to 3.08]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR was defined as the percentage of participants who had a best overall response (BOR) of Complete response (CR), Partial response (PR) or Stable disease (SD) ≥6 weeks prior to any Progressive disease (PD) event and was used to further assess the efficacy of osimertinib compared with SoC EGFR-TKI therapy.
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks until objective disease progression
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Percentage of participants | 97.1 [94.4 to 98.8] | 92.4 [88.6 to 95.2] | 97.2 [90.2 to 99.7] | 95.4 [87.1 to 99.0]
Statistical Analysis 1: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p = 0.0110, Regression, Logistic; Odds Ratio (OR) = 2.78, 95% CI 2-sided [1.25 to 6.78] — An odds ratio > 1 favours osimertinib
Statistical Analysis 2: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.5772, Regression, Logistic; Odds Ratio (OR) = 1.67, 95% CI 2-sided [0.27 to 12.98] — An odds ratio >1 favours osimertinib

6. Secondary Outcome: Depth of Response
Description: The Depth of response was defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions (TLs) at the nadir, in the absence of new lesions (NLs) or progression of Non-target lesions (NTLs), compared to baseline and was used to further assess the efficacy of osimertinib compared with SoC EGFR-TKI therapy
Time Frame: At baseline and every 6 weeks for the first 18 months and then every 12 weeks until objective disease progression
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
percentage of change | -52.36 (25.065) | -45.66 (28.270) | -49.17 (24.303) | -42.92 (26.814)
Statistical Analysis 1: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p = 0.0025, Regression, Linear; Mean Difference (Final Values) = -6.80, 95% CI 2-sided [-11.205 to -2.403]
Statistical Analysis 2: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.1348, Regression, Linear; Mean Difference (Final Values) = -6.59, 95% CI 2-sided [-15.246 to 2.072]

7. Secondary Outcome: Overall Survival (OS)- Number of Participants With an Event
Description: Overall survival was defined as the time from the date of randomisation until death from any cause and was used to further assess the efficacy of osimertinib compared with SoC EGFR-TKI therapy
Time Frame: From first dose to end of study or date of death from any cause, whichever comes first, assessed every 6 weeks (approximately 29 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Participants
  Death | 155 | 166 | 45 | 44
  Still in survival follow-up | 104 | 86 | 25 | 17
  Terminated prior to death | 20 | 25 | 1 | 4
Statistical Analysis 1: Comparison: Osimertinib 80 mg (Global Cohort) vs SoC EGFR-TKI (Global Cohort); Test type: Superiority; p = 0.0462, Log Rank; Hazard Ratio (HR) = 0.799, 95% CI 2-sided [0.6409 to 0.9963]
Statistical Analysis 2: Comparison: Osimertinib 80 mg (China Cohort) vs SoC EGFR-TKI (China Cohort); Test type: Other — The china cohort was not powered for superiority; p = 0.4416, Log Rank; Hazard Ratio (HR) = 0.848, 95% CI 2-sided [0.5568 to 1.2910]

8. Secondary Outcome: Plasma Concentrations of AZD9291
Description: To characterise the pharmacokinetics (PK) of osimertinib
Time Frame: Blood samples collected from each participant at pre-dose, 0.5 to 2 hours, and 3 to 5 hours post-dose on Day 1 Cycle 1, and every other cycle thereafter up to and including Cycle 13 (approximately 9 months)
Population: The pharmacokinetic analysis set (osimertinib arm only) was defined as participants in the FAS who had at least 1 evaluable PK concentration and who had no detectable pre-dose osimertinib concentrations above the lower limit of quantitation (LLQ) on Cycle 1 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nano moles
Arm/Group | Osimertinib 80 mg (Global Cohort) | Osimertinib 80 mg (China Cohort)
Number analyzed (Participants) | 279 | 71
Nano moles
  Cycle 1 Day 1-Predose: number analyzed (Participants) | 199 | 69
  Cycle 1 Day 1-Predose | NA (NA) — NA as values were not calculable and non-quantifiable | NA (NA) — NA as values were not calculable and non-quantifiable
  Cycle 1 Day 1-0.5 - 2 hours: number analyzed (Participants) | 203 | 69
  Cycle 1 Day 1-0.5 - 2 hours | 4.9487 (1173.3679) | 5.0249 (816.7305)
  Cycle 1 Day 1-3 - 5 hours: number analyzed (Participants) | 211 | 69
  Cycle 1 Day 1-3 - 5 hours | 129.3340 (171.2983) | 131.5669 (120.5979)
  Cycle 3 Day 1- Predose: number analyzed (Participants) | 183 | 67
  Cycle 3 Day 1- Predose | 394.3489 (43.9296) | 441.5606 (55.0039)
  Cycle 3 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 183 | 68
  Cycle 3 Day 1, 0.5 - 2 hours | 397.7406 (45.8548) | 441.7343 (60.0626)
  Cycle 3 Day 1, 3 - 5 hours: number analyzed (Participants) | 182 | 67
  Cycle 3 Day 1, 3 - 5 hours | 512.4012 (44.0653) | 553.8090 (60.9883)
  Cycle 5 Day 1, Predose: number analyzed (Participants) | 180 | 67
  Cycle 5 Day 1, Predose | 358.5487 (53.8212) | 419.5893 (63.2507)
  Cycle 5 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 177 | 67
  Cycle 5 Day 1, 0.5 - 2 hours | 369.0696 (51.3284) | 426.8197 (60.3841)
  Cycle 5 Day 1, 3-5 hours: number analyzed (Participants) | 179 | 67
  Cycle 5 Day 1, 3-5 hours | 485.8142 (47.2759) | 570.7729 (61.4401)
  Cycle 7 Day 1-Predose: number analyzed (Participants) | 181 | 62
  Cycle 7 Day 1-Predose | 347.6176 (47.7442) | 397.5857 (54.9006)
  Cycle 7 Day 1-0.5 - 2 hours: number analyzed (Participants) | 179 | 61
  Cycle 7 Day 1-0.5 - 2 hours | 357.8529 (45.0713) | 411.6170 (49.4107)
  Cycle 7 Day 1-3-5 hours: number analyzed (Participants) | 179 | 62
  Cycle 7 Day 1-3-5 hours | 475.6587 (41.5778) | 530.7212 (56.5184)
  Cycle 9 Day 1-Predose: number analyzed (Participants) | 165 | 62
  Cycle 9 Day 1-Predose | 359.5284 (47.0592) | 383.2238 (67.7153)
  Cycle 9 Day 1-0.5-2 hours: number analyzed (Participants) | 165 | 61
  Cycle 9 Day 1-0.5-2 hours | 363.0106 (48.3837) | 395.2179 (71.5532)
  Cycle 9 Day 1-3-5 hours: number analyzed (Participants) | 163 | 62
  Cycle 9 Day 1-3-5 hours | 485.6006 (46.6459) | 490.5964 (70.3383)
  Cycle 11 Day 1-Predose: number analyzed (Participants) | 158 | 59
  Cycle 11 Day 1-Predose | 354.5330 (44.4308) | 410.4023 (66.2329)
  Cycle 11 Day 1-0.5 -2 hours: number analyzed (Participants) | 160 | 59
  Cycle 11 Day 1-0.5 -2 hours | 367.7450 (45.2003) | 415.2427 (64.6174)
  Cycle 11 Day 1-3-5 hours: number analyzed (Participants) | 161 | 59
  Cycle 11 Day 1-3-5 hours | 476.4472 (44.4457) | 528.8081 (68.4645)
  Cycle 13 Day 1-Predose: number analyzed (Participants) | 150 | 55
  Cycle 13 Day 1-Predose | 369.9834 (40.1071) | 404.2678 (62.0291)
  Cycle 13 Day 1-0.5 -2 hours: number analyzed (Participants) | 147 | 54
  Cycle 13 Day 1-0.5 -2 hours | 371.4157 (42.9794) | 393.1688 (62.1053)
  Cycle 13 Day 1-3-5 hours: number analyzed (Participants) | 147 | 55
  Cycle 13 Day 1-3-5 hours | 496.6866 (40.8757) | 499.0220 (62.5485)

9. Secondary Outcome: Plasma Concentrations of Metabolites AZ5104
Description: To characterise the pharmacokinetics (PK) of osimertinib metabolite AZ5104.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nano moles
Arm/Group | Osimertinib 80 mg (Global Cohort) | Osimertinib 80 mg (China Cohort)
Number analyzed (Participants) | 279 | 71
Nano moles
  Cycle 1 Day 1 Predose: number analyzed (Participants) | 207 | 69
  Cycle 1 Day 1 Predose | NA (NA) — NA as the values were non-quantifiable and not calculable | NA (NA) — NA as the values were non-quantifiable and not calculable
  Cycle 1 Day 1-0.5 - 2 hours: number analyzed (Participants) | 207 | 69
  Cycle 1 Day 1-0.5 - 2 hours | 0.1542 (230.5161) | NA (NA) — NA as the values were non-quantifiable and not calculable
  Cycle 1 Day 1-3 - 5 hours: number analyzed (Participants) | 223 | 69
  Cycle 1 Day 1-3 - 5 hours | 3.9399 (153.7651) | 6.3053 (123.9308)
  Cycle 3 Day 1-Predose: number analyzed (Participants) | 183 | 67
  Cycle 3 Day 1-Predose | 42.9123 (50.2410) | 56.8319 (51.0378)
  Cycle 3 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 183 | 68
  Cycle 3 Day 1, 0.5 - 2 hours | 42.7434 (52.8557) | 55.9947 (59.1318)
  Cycle 3 Day 1, 3 - 5 hours: number analyzed (Participants) | 182 | 67
  Cycle 3 Day 1, 3 - 5 hours | 48.3547 (50.4286) | 64.0621 (54.2058)
  Cycle 5 Day 1, Predose: number analyzed (Participants) | 181 | 67
  Cycle 5 Day 1, Predose | 39.3718 (56.6226) | 56.0330 (57.5022)
  Cycle 5 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 178 | 67
  Cycle 5 Day 1, 0.5 - 2 hours | 39.4145 (55.3468) | 55.3767 (55.9096)
  Cycle 5 Day 1, 3-5 hours: number analyzed (Participants) | 180 | 67
  Cycle 5 Day 1, 3-5 hours | 45.6842 (54.3876) | 63.9216 (56.4249)
  Cycle 7 Day 1- Predose: number analyzed (Participants) | 181 | 62
  Cycle 7 Day 1- Predose | 38.3847 (50.0861) | 52.5786 (51.0588)
  Cycle 7 Day 1, 0.5-2 hours: number analyzed (Participants) | 179 | 61
  Cycle 7 Day 1, 0.5-2 hours | 38.5301 (49.6296) | 52.7638 (47.4797)
  Cycle 7 Day 1, 3-5 hours: number analyzed (Participants) | 179 | 62
  Cycle 7 Day 1, 3-5 hours | 44.4670 (48.4730) | 60.6201 (50.6931)
  Cycle 9 Day 1, Predose: number analyzed (Participants) | 165 | 62
  Cycle 9 Day 1, Predose | 40.1230 (47.0682) | 54.4349 (51.3447)
  Cycle 9 Day 1, 0.5-2 hours: number analyzed (Participants) | 165 | 61
  Cycle 9 Day 1, 0.5-2 hours | 40.4987 (47.6483) | 54.7158 (54.6783)
  Cycle 9 Day 1, 3-5 hours: number analyzed (Participants) | 163 | 62
  Cycle 9 Day 1, 3-5 hours | 46.0310 (44.6875) | 60.4649 (52.6147)
  Cycle 11 Day 1, Predose: number analyzed (Participants) | 158 | 59
  Cycle 11 Day 1, Predose | 38.3859 (48.5351) | 56.4782 (59.1303)
  Cycle 11 Day 1, 0.5-2 hours: number analyzed (Participants) | 160 | 59
  Cycle 11 Day 1, 0.5-2 hours | 38.7620 (48.1414) | 57.4095 (57.0891)
  Cycle 11 Day 1, 3-5 hours: number analyzed (Participants) | 161 | 59
  Cycle 11 Day 1, 3-5 hours | 43.9135 (50.6779) | 65.1943 (58.5043)
  Cycle 13 Day 1, Predose: number analyzed (Participants) | 150 | 55
  Cycle 13 Day 1, Predose | 40.4356 (47.2671) | 55.1162 (54.3493)
  Cycle 13 Day 1, 0.5- 2 hours: number analyzed (Participants) | 147 | 54
  Cycle 13 Day 1, 0.5- 2 hours | 40.1116 (46.3929) | 54.3858 (49.9148)
  Cycle 13 Day 1, 3-5 hours: number analyzed (Participants) | 147 | 55
  Cycle 13 Day 1, 3-5 hours | 45.9083 (44.8309) | 61.7426 (51.2924)

10. Secondary Outcome: Plasma Concentrations of Metabolite AZ7550
Description: To characterise the pharmacokinetics (PK) of osimertinib metabolite AZ7550.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nano moles
Arm/Group | Osimertinib 80 mg (Global Cohort) | Osimertinib 80 mg (China Cohort)
Number analyzed (Participants) | 279 | 71
Nano moles
  Cycle 1 Day 1, Predose: number analyzed (Participants) | 207 | 69
  Cycle 1 Day 1, Predose | NA (NA) — NA as the values are not calculable and non-quantifiable. | NA (NA) — NA as the values are not calculable and non-quantifiable.
  Cycle 1 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 207 | 69
  Cycle 1 Day 1, 0.5 - 2 hours | 0.1437 (168.2087) | NA (NA) — NA as the values are not calculable and non-quantifiable.
  Cycle 1 Day 1, 3 - 5 hours: number analyzed (Participants) | 219 | 66
  Cycle 1 Day 1, 3 - 5 hours | 1.8610 (147.4624) | 2.1876 (123.6012)
  Cycle 3 Day 1, Predose: number analyzed (Participants) | 183 | 67
  Cycle 3 Day 1, Predose | 46.1286 (45.1082) | 55.9958 (50.5705)
  Cycle 3 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 183 | 68
  Cycle 3 Day 1, 0.5 - 2 hours | 46.0045 (45.9584) | 55.6754 (53.0925)
  Cycle 3 Day 1, 3 - 5 hours: number analyzed (Participants) | 182 | 67
  Cycle 3 Day 1, 3 - 5 hours | 51.7182 (45.3240) | 62.3493 (53.5513)
  Cycle 5 Day 1, Predose: number analyzed (Participants) | 181 | 67
  Cycle 5 Day 1, Predose | 44.4537 (54.9882) | 53.0434 (52.2936)
  Cycle 5 Day 1, 0.5 - 2 hours: number analyzed (Participants) | 178 | 67
  Cycle 5 Day 1, 0.5 - 2 hours | 45.2186 (51.6418) | 53.1901 (51.5506)
  Cycle 5 Day 1, 3-5 hours: number analyzed (Participants) | 180 | 67
  Cycle 5 Day 1, 3-5 hours | 51.4018 (51.3627) | 62.5218 (51.0627)
  Cycle 7 Day 1, Predose: number analyzed (Participants) | 181 | 62
  Cycle 7 Day 1, Predose | 46.2912 (49.8713) | 53.4167 (50.8399)
  Cycle 7 Day 1, 0.5-2 hours: number analyzed (Participants) | 179 | 61
  Cycle 7 Day 1, 0.5-2 hours | 46.3540 (49.0845) | 54.3942 (46.1253)
  Cycle 7 Day 1,3-5 hours: number analyzed (Participants) | 179 | 62
  Cycle 7 Day 1,3-5 hours | 52.3533 (47.6489) | 61.9004 (51.6117)
  Cycle 9 Day 1, Predose: number analyzed (Participants) | 165 | 62
  Cycle 9 Day 1, Predose | 49.6058 (45.5050) | 54.8207 (50.2534)
  Cycle 9 Day 1, 0.5-2 hours: number analyzed (Participants) | 165 | 61
  Cycle 9 Day 1, 0.5-2 hours | 49.9381 (46.4568) | 55.2437 (52.5736)
  Cycle 9 Day 1, 3-5 hours: number analyzed (Participants) | 163 | 62
  Cycle 9 Day 1, 3-5 hours | 56.5354 (45.6736) | 60.8933 (50.3474)
  Cycle 11 Day 1, Predose: number analyzed (Participants) | 158 | 59
  Cycle 11 Day 1, Predose | 50.9710 (46.8840) | 56.4643 (51.2351)
  Cycle 11 Day 1, 0.5- 2 hours: number analyzed (Participants) | 160 | 59
  Cycle 11 Day 1, 0.5- 2 hours | 51.9773 (45.3186) | 57.4778 (47.3639)
  Cycle 11 Day 1, 3- 5 hours: number analyzed (Participants) | 161 | 59
  Cycle 11 Day 1, 3- 5 hours | 57.6986 (48.2382) | 65.3053 (49.6916)
  Cycle 13 Day 1, Predose: number analyzed (Participants) | 150 | 55
  Cycle 13 Day 1, Predose | 54.5238 (43.8481) | 56.0666 (51.2464)
  Cycle 13 Day 1, 0.5-2 hours: number analyzed (Participants) | 146 | 54
  Cycle 13 Day 1, 0.5-2 hours | 54.1224 (43.7869) | 56.8750 (47.4338)
  Cycle 13 Day 1, 3-5 hours: number analyzed (Participants) | 146 | 55
  Cycle 13 Day 1, 3-5 hours | 61.6053 (42.2947) | 63.3365 (46.3082)

11. Secondary Outcome: Participants Reported Outcome by Cancer Therapy Satisfaction Questionnaire 16 Items (CTSQ-16 Questionnaire)
Description: The CTSQ-16 was a 16-item questionnaire measuring 3 domains related to participant's satisfaction with cancer therapy: Expectations of therapy, Feelings about side effects, and Satisfaction with therapy. Scores ranged from 0 to 100 for each domain, with a higher score associated with the best outcome on each domain. The three domains of interest were separately analysed using an ANCOVA stratified by race (Asian versus Non-Asian) and mutation type (Ex19del versus L858R). The results of the analyses were presented in terms of mean together with standard deviation.
Time Frame: Questionnaire completed in cycle 2 and 3, prior to Week 6 scan (approximately 2 months)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Unit on scale
  Expectations with Therapy, Week 3: number analyzed (Participants) | 227 | 216 | 59 | 60
  Expectations with Therapy, Week 3 | 74.1 (22.42) | 70.3 (21.85) | 77.1 (20.60) | 79.2 (18.58)
  Expectations with Therapy, Week 6: number analyzed (Participants) | 222 | 210 | 60 | 55
  Expectations with Therapy, Week 6 | 76.3 (20.58) | 74.0 (19.46) | 82.2 (17.88) | 82.6 (17.95)
  Feelings about Side-Effects, Week 3: number analyzed (Participants) | 227 | 216 | 59 | 60
  Feelings about Side-Effects, Week 3 | 74.5 (17.22) | 69.1 (20.96) | 73.3 (19.89) | 72.5 (17.46)
  Feelings about Side-Effects, Week 6: number analyzed (Participants) | 222 | 210 | 60 | 55
  Feelings about Side-Effects, Week 6 | 74.6 (19.83) | 69.9 (20.73) | 69.0 (24.46) | 69.7 (20.99)
  Satisfaction with Therapy, Week 3: number analyzed (Participants) | 227 | 216 | 59 | 60
  Satisfaction with Therapy, Week 3 | 84.4 (12.88) | 82.6 (13.60) | 87.2 (12.14) | 86.6 (11.07)
  Satisfaction with Therapy, Week 6: number analyzed (Participants) | 222 | 210 | 60 | 55
  Satisfaction with Therapy, Week 6 | 84.2 (13.94) | 84.6 (12.38) | 87.4 (13.29) | 87.2 (12.06)

12. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life (QLQ) Questionnaires Lung Cancer 13 (QLQ-LC13)
Description: The EORTC QLQ-LC13 was a lung-cancer-specific module comprising 13 questions to assess lung cancer symptoms (cough, haemoptysis, dyspnoea, and site-specific pain); treatment related side-effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia); and pain medication. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items. Higher scores on the global health status/QoL and functioning scales indicated better health status/QoL and function. Higher scores on the symptoms scales indicated greater symptom burden. The analysis was performed using a Mixed-effects model for repeated measures analysis on the change from baseline in PRO symptom score at each visit up to 9 months (281 days), including participants, treatment, visit and treatment by visit interaction as explanatory variables, the baseline PRO score as a covariate along with the baseline PRO score by visit interaction, using an unstructured covariance structure.
Time Frame: Questionnaires completed at baseline, first 9 months, and at week 1, 2, 3, 4, 5, 6, 12, 18, 24, 30 and 36
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Unit on scale
  Dyspnoea, First 9 months: number analyzed (Participants) | 248 | 252 | 67 | 57
  Dyspnoea, First 9 months | -4.04 [-5.63 to -2.45] | -4.14 [-5.73 to -2.54] | -4.87 [-7.81 to -1.92] | -4.82 [-8.01 to -1.63]
  Dyspnoea, week 1: number analyzed (Participants) | 241 | 246 | 67 | 57
  Dyspnoea, week 1 | -3.46 [-5.12 to -1.81] | -3.60 [-5.24 to -1.96] | -1.61 [-5.03 to 1.81] | 0.68 [-3.03 to 4.39]
  Dyspnoea, week 2: number analyzed (Participants) | 236 | 236 | 66 | 57
  Dyspnoea, week 2 | -3.94 [-5.87 to -2.00] | -3.64 [-5.57 to -1.70] | -2.27 [-6.01 to 1.48] | -5.03 [-9.08 to -0.98]
  Dyspnoea, week 3: number analyzed (Participants) | 239 | 237 | 63 | 57
  Dyspnoea, week 3 | -3.99 [-5.85 to -2.12] | -3.27 [-5.14 to -1.41] | -3.09 [-6.96 to 0.77] | -5.55 [-9.69 to -1.42]
  Dyspnoea, week 4: number analyzed (Participants) | 206 | 211 | 63 | 53
  Dyspnoea, week 4 | -4.81 [-6.59 to -3.02] | -4.11 [-5.88 to -2.34] | -5.35 [-8.72 to -1.99] | -5.55 [-9.20 to -1.89]
  Dyspnoea, week 5: number analyzed (Participants) | 199 | 196 | 57 | 55
  Dyspnoea, week 5 | -3.51 [-5.53 to -1.50] | -5.19 [-7.22 to -3.17] | -5.72 [-10.06 to -1.39] | -5.76 [-10.32 to -1.20]
  Dyspnoea, week 6: number analyzed (Participants) | 222 | 214 | 64 | 53
  Dyspnoea, week 6 | -4.51 [-6.47 to -2.56] | -4.45 [-6.42 to -2.48] | -4.83 [-8.53 to -1.12] | -6.37 [-10.40 to -2.33]
  Dyspnoea, week 12: number analyzed (Participants) | 225 | 203 | 61 | 52
  Dyspnoea, week 12 | -3.83 [-5.99 to -1.68] | -5.75 [-7.96 to -3.54] | -5.38 [-9.41 to -1.35] | -6.67 [-11.04 to -2.30]
  Dyspnoea, week 18: number analyzed (Participants) | 214 | 199 | 59 | 52
  Dyspnoea, week 18 | -4.97 [-7.18 to -2.76] | -5.21 [-7.46 to -2.95] | -7.67 [-11.54 to -3.79] | -7.48 [-11.66 to -3.30]
  Dyspnoea, week 24: number analyzed (Participants) | 202 | 185 | 55 | 47
  Dyspnoea, week 24 | -4.65 [-7.06 to -2.25] | -4.56 [-7.02 to -2.09] | -7.59 [-11.84 to -3.34] | -5.67 [-10.27 to -1.08]
  Dyspnoea, week 30: number analyzed (Participants) | 195 | 172 | 55 | 49
  Dyspnoea, week 30 | -3.89 [-6.34 to -1.45] | -3.68 [-6.22 to -1.15] | -5.81 [-10.59 to -1.02] | -3.46 [-8.58 to 1.65]
  Dyspnoea, week 36: number analyzed (Participants) | 184 | 151 | 52 | 43
  Dyspnoea, week 36 | -2.88 [-5.52 to -0.24] | -2.04 [-4.83 to 0.75] | -4.21 [-8.91 to 0.48] | -2.18 [-7.28 to 2.93]
  Cough, First 9 months: number analyzed (Participants) | 248 | 252 | 67 | 57
  Cough, First 9 months | -10.97 [-12.77 to -9.17] | -11.65 [-13.47 to -9.84] | -13.75 [-17.17 to -10.33] | -8.49 [-12.19 to -4.79]
  Cough, week 1: number analyzed (Participants) | 241 | 246 | 67 | 57
  Cough, week 1 | -6.90 [-9.30 to -4.51] | -4.83 [-7.20 to -2.46] | -4.60 [-9.00 to -0.20] | -3.69 [-8.46 to 1.07]
  Cough, week 2: number analyzed (Participants) | 236 | 236 | 66 | 57
  Cough, week 2 | -9.04 [-11.58 to -6.49] | -9.52 [-12.05 to -6.98] | -12.26 [-17.15 to -7.37] | -3.73 [-9.01 to 1.54]
  Cough, week 3: number analyzed (Participants) | 239 | 237 | 63 | 57
  Cough, week 3 | -9.78 [-12.37 to -7.20] | -10.24 [-12.82 to -7.65] | -11.95 [-16.66 to -7.24] | -5.56 [-10.57 to -0.54]
  Cough, week 4: number analyzed (Participants) | 206 | 211 | 63 | 53
  Cough, week 4 | -11.25 [-13.87 to -8.63] | -13.36 [-15.96 to -10.76] | -12.78 [-17.80 to -7.77] | -10.32 [-15.75 to -4.90]
  Cough, week 5: number analyzed (Participants) | 199 | 196 | 57 | 55
  Cough, week 5 | -12.98 [-15.64 to -10.31] | -13.55 [-16.21 to -10.88] | -17.74 [-23.11 to -12.38] | -9.20 [-14.84 to -3.55]
  Cough, week 6: number analyzed (Participants) | 222 | 214 | 64 | 53
  Cough, week 6 | -11.88 [-14.56 to -9.19] | -11.92 [-14.63 to -9.21] | -16.92 [-22.36 to -11.48] | -10.58 [-16.52 to -4.64]
  Cough, week 12: number analyzed (Participants) | 225 | 203 | 61 | 52
  Cough, week 12 | -13.36 [-15.95 to -10.78] | -13.57 [-16.24 to -10.90] | -15.51 [-21.39 to -9.64] | -8.04 [-14.41 to -1.67]
  Cough, week 18: number analyzed (Participants) | 214 | 199 | 59 | 52
  Cough, week 18 | -12.31 [-15.25 to -9.37] | -11.00 [-14.03 to -7.98] | -11.79 [-17.19 to -6.40] | -9.44 [-15.23 to -3.65]
  Cough, week 24: number analyzed (Participants) | 202 | 185 | 55 | 47
  Cough, week 24 | -11.34 [-14.24 to -8.43] | -13.16 [-16.17 to -10.14] | -17.61 [-22.84 to -12.39] | -14.92 [-20.56 to -9.29]
  Cough, week 30: number analyzed (Participants) | 195 | 172 | 55 | 49
  Cough, week 30 | -10.34 [-13.21 to -7.46] | -12.43 [-15.44 to -9.41] | -15.45 [-21.46 to -9.45] | -9.35 [-15.75 to -2.94]
  Cough, week 36: number analyzed (Participants) | 184 | 151 | 52 | 43
  Cough, week 36 | -11.49 [-14.48 to -8.49] | -14.62 [-17.85 to -11.39] | -14.62 [-20.65 to -8.58] | -8.55 [-15.14 to -1.96]
  Pain in Chest, First 9 months: number analyzed (Participants) | 248 | 252 | 67 | 57
  Pain in Chest, First 9 months | -6.62 [-8.24 to -5.01] | -6.41 [-8.04 to -4.78] | -2.79 [-5.84 to 0.26] | -4.74 [-8.05 to -1.44]
  Pain in Chest, week 1: number analyzed (Participants) | 241 | 246 | 67 | 57
  Pain in Chest, week 1 | -1.93 [-4.19 to 0.32] | -4.26 [-6.50 to -2.03] | -1.79 [-5.98 to 2.40] | -4.16 [-8.71 to 0.38]
  Pain in Chest, week 2: number analyzed (Participants) | 236 | 236 | 66 | 57
  Pain in Chest, week 2 | -5.94 [-8.13 to -3.74] | -6.32 [-8.51 to -4.13] | -4.76 [-8.63 to -0.89] | -3.00 [-7.18 to 1.17]
  Pain in Chest, week 3: number analyzed (Participants) | 239 | 237 | 63 | 57
  Pain in Chest, week 3 | -7.17 [-9.31 to -5.04] | -5.36 [-7.49 to -3.23] | -0.76 [-4.90 to 3.39] | -4.77 [-9.18 to -0.36]
  Pain in Chest, week 4: number analyzed (Participants) | 206 | 211 | 63 | 53
  Pain in Chest, week 4 | -7.45 [-9.60 to -5.29] | -6.40 [-8.54 to -4.26] | -2.13 [-6.32 to 2.07] | -4.22 [-8.78 to 0.34]
  Pain in Chest, week 5: number analyzed (Participants) | 199 | 196 | 57 | 55
  Pain in Chest, week 5 | -7.33 [-9.54 to -5.11] | -6.98 [-9.20 to -4.76] | -0.62 [-4.67 to 3.42] | -6.82 [-11.05 to -2.60]
  Pain in Chest, week 6: number analyzed (Participants) | 222 | 214 | 64 | 53
  Pain in Chest, week 6 | -4.99 [-7.30 to -2.68] | -7.08 [-9.41 to -4.75] | 0.94 [-3.40 to 5.29] | -6.26 [-11.00 to -1.52]
  Pain in Chest, week 12: number analyzed (Participants) | 225 | 203 | 61 | 52
  Pain in Chest, week 12 | -7.28 [-9.56 to -5.01] | -6.70 [-9.05 to -4.35] | -3.71 [-8.77 to 1.35] | -5.13 [-10.62 to 0.36]
  Pain in Chest, week 18: number analyzed (Participants) | 214 | 199 | 59 | 52
  Pain in Chest, week 18 | -6.79 [-9.22 to -4.36] | -7.90 [-10.40 to -5.41] | -4.40 [-9.05 to 0.26] | -7.24 [-12.23 to -2.25]
  Pain in Chest, week 24: number analyzed (Participants) | 202 | 185 | 55 | 47
  Pain in Chest, week 24 | -7.72 [-10.26 to -5.18] | -7.34 [-9.95 to -4.72] | -5.66 [-10.48 to -0.84] | -3.15 [-8.36 to 2.07]
  Pain in Chest, week 30: number analyzed (Participants) | 195 | 172 | 55 | 49
  Pain in Chest, week 30 | -8.33 [-10.80 to -5.87] | -6.60 [-9.18 to -4.02] | -4.25 [-9.62 to 1.12] | -4.02 [-9.76 to 1.72]
  Pain in Chest, week 36: number analyzed (Participants) | 184 | 151 | 52 | 43
  Pain in Chest, week 36 | -7.94 [-10.59 to -5.30] | -5.58 [-8.43 to -2.73] | -3.56 [-9.42 to 2.30] | -3.40 [-9.80 to 3.00]

13. Secondary Outcome: Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 Items (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 cancer-specific questionnaire consisted of 30 questions, combined to produce 5 functional scales, 3 symptom scales, 6 individual items, and a global measure of health status/QoL. An outcome variable consisting of a score from 0 to 100 was derived for each of the symptom scales/symptom items, the functional scales, and the global health status/QoL scale in the EORTC QLQ-C30. Higher scores on the global health status and functioning scales indicated better health status/function. Higher scores on the symptoms scales indicated greater symptom burden. The analysis was performed using a Mixed-effects model for repeated measures analysis on the change from baseline in PRO symptom score at each visit up to 9 months (281 days), including participants, treatment, visit and treatment by visit interaction as explanatory variables, the baseline PRO score as a covariate along with the baseline PRO score by visit interaction, using an unstructured covariance structure.
Time Frame: Questionnaires completed at baseline, first 9 months, and at week 6, 12, 18, 24, 30, and 36.
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Unit on scale
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
Number analyzed (Participants) | 279 | 277 | 71 | 65
Unit on scale
  Fatigue, First 9 months: number analyzed (Participants) | 252 | 247 | 68 | 63
  Fatigue, First 9 months | -5.48 [-7.45 to -3.52] | -4.72 [-6.74 to -2.69] | -5.65 [-9.33 to -1.98] | -5.79 [-9.58 to -2.00]
  Fatigue, week 6: number analyzed (Participants) | 239 | 236 | 68 | 63
  Fatigue, week 6 | -4.13 [-6.35 to -1.91] | -5.78 [-8.02 to -3.54] | -1.73 [-6.05 to 2.58] | -6.81 [-11.30 to -2.33]
  Fatigue, week 12: number analyzed (Participants) | 237 | 210 | 65 | 61
  Fatigue, week 12 | -5.11 [-7.31 to -2.91] | -6.52 [-8.81 to -4.23] | -5.40 [-9.51 to -1.29] | -6.36 [-10.61 to -2.12]
  Fatigue, week 18: number analyzed (Participants) | 229 | 214 | 61 | 60
  Fatigue, week 18 | -6.83 [-9.21 to -4.44] | -5.77 [-8.23 to -3.31] | -6.64 [-11.26 to -2.03] | -7.90 [-12.61 to -3.19]
  Fatigue, week 24: number analyzed (Participants) | 216 | 195 | 57 | 57
  Fatigue, week 24 | -6.18 [-8.75 to -3.61] | -4.96 [-7.63 to -2.28] | -8.92 [-13.30 to -4.54] | -3.87 [-8.32 to 0.58]
  Fatigue, week 30: number analyzed (Participants) | 207 | 178 | 57 | 56
  Fatigue, week 30 | -5.19 [-7.94 to -2.43] | -3.26 [-6.16 to -0.35] | -4.43 [-9.53 to 0.68] | -6.31 [-11.53 to -1.10]
  Fatigue, week 36: number analyzed (Participants) | 193 | 158 | 55 | 50
  Fatigue, week 36 | -5.47 [-8.31 to -2.63] | -2.00 [-2.00 to 1.04] | -6.78 [-12.38 to -1.19] | -3.46 [-9.28 to 2.36]
  Appetite Loss, First 9 months: number analyzed (Participants) | 252 | 247 | 68 | 63
  Appetite Loss, First 9 months | -6.15 [-8.39 to -3.90] | -5.64 [-7.96 to -3.32] | 1.18 [-2.78 to 5.14] | -1.73 [-5.80 to 2.34]
  Appetite Loss, week 6: number analyzed (Participants) | 239 | 236 | 68 | 63
  Appetite Loss, week 6 | -4.54 [-7.36 to -1.72] | -5.67 [-8.52 to -2.83] | 3.20 [-1.60 to 8.01] | -6.27 [-11.26 to -1.27]
  Appetite Loss, week 12: number analyzed (Participants) | 237 | 210 | 65 | 61
  Appetite Loss, week 12 | -6.52 [-9.43 to -3.62] | -6.95 [-9.98 to -3.91] | 1.58 [-3.23 to 6.39] | -1.44 [-6.41 to 3.53]
  Appetite Loss, week 18: number analyzed (Participants) | 229 | 214 | 61 | 60
  Appetite Loss, week 18 | -7.27 [-10.09 to -4.45] | -6.84 [-9.75 to -3.92] | 1.42 [-4.38 to 7.22] | -4.43 [-10.35 to 1.48]
  Appetite Loss, week 24: number analyzed (Participants) | 216 | 195 | 57 | 57
  Appetite Loss, week 24 | -7.14 [-10.27 to -4.01] | -5.08 [-8.35 to -1.81] | -2.26 [-7.74 to 3.22] | 0.24 [-5.29 to 5.78]
  Appetite Loss, week 30: number analyzed (Participants) | 207 | 178 | 57 | 56
  Appetite Loss, week 30 | -4.50 [-7.74 to -1.26] | -4.17 [-7.60 to -0.74] | 2.19 [-3.28 to 7.65] | -1.83 [-7.36 to 3.70]
  Appetite Loss, week 36: number analyzed (Participants) | 193 | 158 | 55 | 50
  Appetite Loss, week 36 | -6.90 [-10.00 to -3.81] | -5.15 [-8.49 to -1.81] | 0.98 [-5.28 to 7.24] | 3.36 [-3.15 to 9.86]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from the time of signature of informed consent throughout the Treatment Period and including the safety follow-up period.The safety follow-up period was defined as 28 days after study drug was discontinued
Description: An adverse event was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. In clinical studies, an AE included an undesirable medical condition occurring at any time, including run-in or washout periods, even if no study treatment had been administered. The term AE was used to include both serious and non-serious AEs.
Arm/Group | Osimertinib 80 mg (Global Cohort) | SoC EGFR-TKI (Global Cohort) | Osimertinib 80 mg (China Cohort) | SoC EGFR-TKI (China Cohort)
All-Cause Mortality (participants affected / at risk) | 155/279 | 166/277 | 45/71 | 44/65
Serious Adverse Events (participants affected / at risk) | 74/279 | 76/277 | 25/71 | 12/65
Other Adverse Events (participants affected / at risk) | 273/279 | 271/277 | 70/71 | 64/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib 80 mg (Global Cohort) (N=279) | SoC EGFR-TKI (Global Cohort) (N=277) | Osimertinib 80 mg (China Cohort) (N=71) | SoC EGFR-TKI (China Cohort) (N=65)
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 2 | 0 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Empyema (Infections and infestations) | 1 | 0 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0 | 0
Pleural infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 7 | 3 | 1
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 0 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Salmonella bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Histiocytic necrotising lymphadenitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Aortic dissection (Vascular disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 0
Embolism (Vascular disorders) | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 5 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 3 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Asthenia (General disorders) | 2 | 2 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Condition aggravated (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 1 | 1 | 0
Drug withdrawal syndrome (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Adenoviral upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Cerebral ventricle dilatation (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Hepatitis C (Hepatobiliary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Osimertinib 80 mg (Global Cohort) (N=279) | SoC EGFR-TKI (Global Cohort) (N=277) | Osimertinib 80 mg (China Cohort) (N=71) | SoC EGFR-TKI (China Cohort) (N=65)
Diarrhoea (Gastrointestinal disorders) | 167 | 162 | 17 | 19
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 73 | 136 | 14 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 92 | 92 | 4 | 8
Paronychia (Infections and infestations) | 89 | 84 | 9 | 2
Stomatitis (Gastrointestinal disorders) | 82 | 60 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 66 | 58 | 10 | 8
Aspartate aminotransferase increased (Investigations) | 28 | 69 | 11 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 50 | 44 | 5 | 4
Nausea (Gastrointestinal disorders) | 55 | 55 | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 60 | 50 | 14 | 11
Constipation (Gastrointestinal disorders) | 51 | 39 | 4 | 3
Fatigue (General disorders) | 45 | 35 | 7 | 6
Vomiting (Gastrointestinal disorders) | 41 | 32 | 10 | 5
Anaemia (Blood and lymphatic system disorders) | 44 | 27 | 27 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 42 | 22 | 10 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 35 | 1 | 5
Headache (Nervous system disorders) | 39 | 25 | 7 | 4
Alanine aminotransferase increased (Investigations) | 19 | 74 | 6 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 29 | 7 | 6
Insomnia (Psychiatric disorders) | 31 | 21 | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 36 | 23 | 9 | 3
Electrocardiogram QT prolonged (Investigations) | 28 | 12 | 6 | 3
Pyrexia (General disorders) | 32 | 12 | 0 | 0
Dry eye (Eye disorders) | 21 | 21 | 0 | 0
Oedema peripheral (General disorders) | 16 | 24 | 0 | 0
Conjunctivitis (Infections and infestations) | 18 | 21 | 1 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 21 | 0 | 0
Dysgeusia (Nervous system disorders) | 18 | 9 | 0 | 0
Asthenia (General disorders) | 27 | 10 | 5 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 28 | 14 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 14 | 0 | 0
Weight decreased (Investigations) | 20 | 20 | 17 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 19 | 14 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 18 | 16 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 13 | 19 | 12 | 8
White blood cell count decreased (Investigations) | 27 | 5 | 29 | 6
Dizziness (Nervous system disorders) | 22 | 13 | 3 | 4
Pneumonia (Infections and infestations) | 24 | 11 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 24 | 13 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 14 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 0 | 7 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 15 | 12 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 12 | 15 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 18 | 10 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 17 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 21 | 3 | 12 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 | 6 | 7 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 16 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 21 | 1 | 12 | 2
Blood alkaline phosphatase increased (Investigations) | 7 | 15 | 6 | 4
Platelet count decreased (Investigations) | 15 | 4 | 20 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 17 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 12 | 6
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 12 | 7
Proteinuria (Renal and urinary disorders) | 0 | 0 | 9 | 7
Urinary tract infection (Infections and infestations) | 17 | 12 | 8 | 8
Lymphocyte count decreased (Investigations) | 0 | 0 | 11 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 7 | 7
Chest discomfort (General disorders) | 0 | 0 | 6 | 8
Non-cardiac chest pain (General disorders) | 18 | 17 | 8 | 5
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 6 | 7
Haematuria (Renal and urinary disorders) | 0 | 0 | 8 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 17 | 10 | 9 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 3 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 5 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 3
Hypertension (Vascular disorders) | 15 | 10 | 4 | 5
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 2 | 5
Blood creatinine increased (Investigations) | 0 | 0 | 5 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 5 | 2
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 2
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 5 | 4
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 2 | 5
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 2 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 2
Haemoglobin decreased (Investigations) | 0 | 0 | 2 | 4
Blood uric acid increased (Investigations) | 0 | 0 | 4 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 38 | 46 | 10 | 12

LIMITATIONS AND CAVEATS:
There were 19 Chinese participants who were included in both the global and China cohort which gives a total of 692 participants instead of a total of 673 participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT02296125/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/25/NCT02296125/SAP_001.pdf